CLINICAL TRIAL: NCT06664372
Title: Insertion of Frontal Ventricular Catheter of VP Shunt in Congenital Hydrocephalus Guided by Trans Fontanelle Ultrasound
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Salah Mohamed Omran, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Transfontanelle US vp shunt
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Ventriculoperitoneal Shunt; Trans Fontanelle US; Congenital Hydrocephalus
Keywords: ventriculoperitoneal shunt; Trans fontanelle US; Congenital hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Trans fontanelle US Guided VP Shunt (Experimental): insertion of proximal vp shunt by trans fontanelle US
  Interventions: Procedure: Trans fontanelle US Guided VP Shunt

INTERVENTIONS:
Procedure: Trans fontanelle US Guided VP Shunt — Insertion of proximal VP shunt catheter by trans fontanelle US

SUMMARY:
The Aim of This Study Is To Evaluate The Role Of Ultrasound In Decreasing Rate Of Proximal Obstruction In Frontal VP Shunt

DETAILED DESCRIPTION:
Congenital Hydrocephalus is a very common congenital anomalie known as the abnormal accumulation of csf in the ventricles and subarachnoid spaces under high tension due to imbalance between synthesis and absorption of csf , The incidence of congenital hydrocephalus is higher in low income country than in high income countries Treatment options for hydrocephalus are multiple but the most common treatment option world wide is VP Shunt . Although, VP Shunt still has a high rate of failure as revisions are required in 30% - 40% of cases In Vp shunt insertion , the placement of ventricular catheter is done mainly by free hand technique but recently The trans fontanelle ultrasound guided placement of ventricular catheter become a standard technique in multiple centers The free hand technique has low accuracy rate in proper intraventricular placement of the proximal catheter than the ultrasound guided technique . On the other hand , the use of intra operative ultrasound can visualize the anatomy of lateral ventricles and choroid plexus which makes the placement of ventricular catheter more accurate than the blind free hand technique So we are aiming in this study to highlight the efficacy of ultrasound guided placement of ventricular catheter of the frontal shunt in decreasing the rate of proximal catheter obstruction and we choose the frontal shunt because it has an advantage over the occipital in rate of revisions as it has a lower rate

ELIGIBILITY:
Inclusion Criteria:

* patients who are diagnosed with congenital Hydrocephalus
* age of patients : < 2 years with patent Anterior Fontanelle
* Not operated with frontal shunt before

Exclusion Criteria:

* patients who are diagnosed with congenital Hydrocephalus
* age of patients : < 2 years with patent Anterior Fontanelle
* Not operated with frontal shunt before

Ages: 5 Days to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate Of Proximal Revisions In Frontal Shunt | 2 years

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang Z, Zhang Y, Hu F, Ding J, Wang X. Pathogenesis and pathophysiology of idiopathic normal pressure hydrocephalus. CNS Neurosci Ther. 2020 Dec;26(12):1230-1240. doi: 10.1111/cns.13526. Epub 2020 Nov 26. PMID 33242372
- [Background] Sarikaya-Seiwert S, Schievelkamp AH, Born M, Wispel C, Haberl H, Shabo E. The impact of real-time ultrasound guidance on ventricular catheter placement in cerebrospinal fluid shunts - a single-center study. Ultraschall Med. 2025 Apr;46(2):170-176. doi: 10.1055/a-2352-9404. Epub 2024 Jun 25. PMID 38917967
- [Background] Kullmann M, Khachatryan M, Schuhmann MU. Ultrasound-guided placement of ventricular catheters in first-time pediatric VP shunt surgery. Childs Nerv Syst. 2018 Mar;34(3):465-471. doi: 10.1007/s00381-017-3660-2. Epub 2017 Nov 22. PMID 29167995